CLINICAL TRIAL: NCT01157169
Title: A Single-Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalence Study of Buprenorphine 8 mg Sublingual Tablets Under Fasting Conditions.
Brief Title: Buprenorphine 8 mg Sublingual Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: TEVA Pharmaceuticals, USA
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-A63-AU
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Results first posted 2010-09-13 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Test Product (Experimental): Buprenorphine 8 mg Sublingual Tablets
  Interventions: Drug: Buprenorphine
- Reference Listed Drug (Active Comparator): Subutex® 8 mg Sublingual Tablets
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — 8 mg Sublingual Tablets
  Arms: Investigational Test Product
Drug: Buprenorphine — 8 mg Sublingual Tablets
  Other Names: Subutex®
  Arms: Reference Listed Drug

SUMMARY:
The object of this study is to compare the rate and extent of absorption of an investigational formulation of buprenorphine 8 mg sublingual tablets manufactured by Barr Laboratories, Inc. to an equivalent oral dose of the commercially available reference product, Subutex® manufactured by Reckitt Benckiser, following and overnight fast of at least 10 hours.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a male or non-pregnant, non-breastfeeding female.
* Subject must be between 18 and 45 years of age (inclusive).
* Subject's Body Mass Index (BMI) must be between 18 and 30 (inclusive), and subject must weigh a minimum of 50 kg (110 lbs).
* Female subjects must agree to utilize one of the following forms of contraception from screening through 4 weeks after completion of the study. Approved forms of contraception are abstinence, double barrier, IUD in place at least 30 days prior to study drug administration, vasectomized partner, surgically sterile for at least 6 months, or at least 2 years postmenopausal.
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to completion of any study-specific procedures.
* Subject is willing and able to remain in the study unit for the entire duration of the confinement period and return for all scheduled outpatient visits.

Exclusion Criteria:

* History or presence of any clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results.
* History or presence of pancreatitis, bowel obstruction, glaucoma, enlargement of the prostate, adrenal disease, hyperthyroidism, or gallbladder disease. Subjects with a history of cholecystectomy for the treatment of gallbladder disease will be excluded.
* Females taking any oral contraceptives including estrogen and progestin combined pills, progestin-only pills, patch, or vaginal ring within 28 days prior to the first dose of study medication; using injectable contraceptives within 6 months of first dose; or who have ever had progestational hormone implants.
* Females taking hormone replacement therapy within 60 days prior to the first dose of study medication.
* Has a clinically significant abnormal finding on the physical exam, medical history, ECG, or clinical laboratory results at screening.
* History or presence of allergic or adverse response to buprenorphine, naltrexone, or any comparable or similar product.
* Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in another clinical trial within 30 days prior to the first dose of study medication.
* Has used any over-the-counter (OTC) medication, including cough and cold preparations, vitamins, and herbal supplements, within 7 days prior to the first dose of study medication.
* Has used any prescription medication within 14 days prior to the first dose of study medication.
* Has consumed beverages or food containing alcohol, caffeine/xanthine, or poppy seeds from 48 hours prior to the first dose of study medication or has consumed beverages or foods containing grapefruit from 14 days prior to the first dose of study medication.
* Has been treated with any known enzyme-altering drugs, such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication.
* Has smoked or used tobacco products within 60 days prior to the first dose of study medication.
* Has a history of treatment for substance abuse (including alcohol) in the past 5 years.
* Is a female with a positive pregnancy test result.
* Has any piercing of the tongue or has a lip piercing within 30 days prior to the first dose of study medication.
* Has a positive urine screen for drugs of abuse.
* Has a positive urine alcohol test or ethanol breath test.
* Has a positive test for or has been treated for hepatitis B, hepatitis C, or HIV.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A Bieberdorf, M.D., CPI, Principal Investigator — CEDRA Clinical Research, LLC
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine (Test) First: 8 mg Buprenorphine Sublingual Tablets test product dosed in first period followed by 8 mg Subutex® Sublingual Tablets reference product dosed in the second period.
- Subutex® (Reference) First: 8 mg Subutex® Sublingual Tablets reference product dosed in first period followed by 8 mg Buprenorphine Sublingual Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Buprenorphine (Test) First | Subutex® (Reference) First
Started | 20 | 20
Completed | 16 | 18
Not Completed | 4 | 2
Not completed — Emesis Within 4 hrs of Administration | 4 | 2
Period: Washout of 10 Days
Arm/Group | Buprenorphine (Test) First | Subutex® (Reference) First
Started | 16 | 18
Completed | 16 | 18
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Buprenorphine (Test) First | Subutex® (Reference) First
Started | 16 | 18
Completed | 16 | 17
Not Completed | 0 | 1
Not completed — Emesis Within 4 hrs of Administration | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine (Test) First | Subutex® (Reference) First | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 11 | 14 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 2
  Black | 3 | 1 | 4
  Caucasian | 9 | 12 | 21
  Hispanic | 7 | 5 | 12
  American Indian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Buprenorphine.
Description: Bioequivalence based on Buprenorphine Cmax (maximum observed concentration of drug substance in plasma).
Time Frame: Blood samples collected over a 144 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Buprenorphine (Test): 8 mg Buprenorphine Sublingual Tablets test product dosed in either period.
- Subutex® (Reference): 8 mg Subutex® Sublingual Tablets reference product dosed in either period.
Arm/Group | Buprenorphine (Test) | Subutex® (Reference)
Number analyzed (Participants) | 33 | 33
ng/mL | 4.40 (2.16) | 3.88 (1.82)
Statistical Analysis 1: Comparison: Buprenorphine (Test) vs Subutex® (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 110.49, 90% CI 2-sided [101.67 to 120.07] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t for Buprenorphine.
Description: Bioequivalence based on Buprenorphine AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration).
Time Frame: Blood samples collected over a 144 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Buprenorphine (Test) | Subutex® (Reference)
Number analyzed (Participants) | 33 | 33
ng*h/mL | 35.12 (12.55) | 32.92 (12.04)
Statistical Analysis 1: Comparison: Buprenorphine (Test) vs Subutex® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 105.91, 90% CI 2-sided [99.74 to 112.45] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf for Buprenorphine.
Description: Bioequivalence based on Buprenorphine AUC0-inf (area under the concentration-time curve from time zero to infinity).
Time Frame: Blood samples collected over a 144 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Buprenorphine (Test) | Subutex® (Reference)
Number analyzed (Participants) | 33 | 33
ng*h/mL | 37.19 (13.39) | 35.73 (13.93)
Statistical Analysis 1: Comparison: Buprenorphine (Test) vs Subutex® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 103.97, 90% CI 2-sided [97.18 to 111.24] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Cmax for Norbuprenorphine.
Description: Informational comparison of Cmax (maximum observed concentration of drug substance in plasma) values for the metabolite Norbuprenorphine.
Time Frame: Blood samples collected over a 144 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Buprenorphine (Test) | Subutex® (Reference)
Number analyzed (Participants) | 33 | 33
ng/mL | 1.58 (0.719) | 1.64 (0.643)
Statistical Analysis 1: Comparison: Buprenorphine (Test) vs Subutex® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 93.28, 90% CI 2-sided [85.37 to 101.93] — This analysis was for informational purposes only and was not used to establish bioequivalence

5. Secondary Outcome: AUC0-t for Norbuprenorphine.
Description: Informational comparison of AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration) values for the metabolite Norbuprenorphine.
Time Frame: Blood samples collected over a 144 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Buprenorphine (Test) | Subutex® (Reference)
Number analyzed (Participants) | 33 | 33
ng*h/mL | 45.34 (18.72) | 47.58 (17.91)
Statistical Analysis 1: Comparison: Buprenorphine (Test) vs Subutex® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 94.19, 90% CI 2-sided [87.44 to 101.46] — This analysis was for informational purposes only and was not used to establish bioequivalence

6. Secondary Outcome: AUC0-inf for Norbuprenorphine.
Description: Informational comparison of AUC0-inf (area under the concentration-time curve from time zero to infinity) values for the metabolite Norbuprenorphine.
Time Frame: Blood samples collected over a 144 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Buprenorphine (Test) | Subutex® (Reference)
Number analyzed (Participants) | 33 | 33
ng*h/mL | 50.77 (28.99) | 51.04 (22.12)
Statistical Analysis 1: Comparison: Buprenorphine (Test) vs Subutex® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 95.06, 90% CI 2-sided [86.56 to 104.39] — This analysis was for informational purposes only and was not used to establish bioequivalence

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 3 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Buprenorphine (Test) First | Subutex® (Reference) First
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 22/40 | 13/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine (Test) First (N=40) | Subutex® (Reference) First (N=40)
Nausea (General disorders) | 15 (15) | 8 (8)
Dizziness (General disorders) | 8 (8) | 3 (3)
Headache (General disorders) | 6 (6) | 6 (6)
Emesis (General disorders) | 9 (9) | 3 (3)
Fatigue (General disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.